CLINICAL TRIAL: NCT02634918
Title: Ultrasonography in Hemophilic Joint Disease
Brief Title: Ultrasonography in Hemophilic Joint Disease and Serum Markers
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Suchitra Acharya, Professor of Pediatrics, Northwell Health
Other Study IDs: #15-145
Record Dates: First submitted 2015-10-08; First posted 2015-12-18 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Hemophilia A; Hemophilia B; Hemarthroses
Keywords: ultrasound,; ultrasonography; hemophilic joint; Doppler
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Hemarthrosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples for angiogenic and cartilage degradation markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ultrasound: 3 groups of hemophilia patients - Those with > 20 bleeds into a joint, those with < 2 bleeds into a joint and those with no bleeds into a joint will be enrolled into the study
  Interventions: Other: ultrasound
- those with < 2 bleeds into a joint and: 3 groups of hemophilia patients Group I - Those with > 20 bleeds into a joint, Group II - those with < 2 bleeds into a joint and Group III - those with no bleeds into a joint will be enrolled into the study
  Interventions: Other: ultrasound
- those with no bleeds into a joint will be enrolled into the st: 3 groups of hemophilia patients Group I - Those with > 20 bleeds into a joint, Group II - those with < 2 bleeds into a joint and Group III - those with no bleeds into a joint will be enrolled into the study
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — ultrasound will be performed in hemophilia boys with a history of 20 joint bleeds- Group I, less than 2 joint bleeds into a joint -Group II and no joint bleeds- Group III

SUMMARY:
Hemophilia is a bleeding disorder (deficiency of a blood clotting factor/ protein) resulting in bleeding in joints and muscles. As patients continue to bleed into their joints they develop progressive joint damage leading to joint contractures, disability and days missed from work and school resulting in chronic debilitating pain and compromised quality of life. Current therapy is the administration of the missing protein or factor concentrate on a scheduled basis to prevent bleeding into the joints referred to as prophylaxis. This factor concentrate is expensive ~ $ 3,000 - 6,000 per infusion/ week in a child weighing 20 kg translating into $ 77,000 /yr for life. This regimen has been shown to be effective to prevent joint bleeds but the timing is unclear and not based on adequate evidence. Currently joint damage is diagnosed using MRI which is expensive and requires sedation in children < 6 yrs of age. Therefore there is a need for a user friendly tool such as a ultrasound to monitor for the development of joint disease and tailor treatment based on an individual child's needs. This would also enable differentiating a joint bleed from a soft tissue bleed which present similarly and duration of treatment tends to be longer for a joint bleed. Acharya et al have previously shown that ultrasound is comparable to MRI for the diagnosis of hemophilic joint disease in hemophilia patients over the age of 6 years. However, the diagnostic findings in children < 18 years with hemophilia on ultrasound is not well defined(1).

The hemophilic synovium after repeated joint bleeds reveals the development of new vessels which are fragile and contribute to recurrent joint bleeds. Acharya et al have previously shown that angiogenesis, a process of new vessel formation is active in hemophilic synovium and angiogenic markers were significantly elevated in hemophilic patients with joint disease when compared to those without (2). Since ultrasound can detect these new vessel changes in the hemophilic synovium in hemophilia patients with joint disease and hemophilia patients with joint disease demonstrate elevated markers of new vessel formation these investigators would now like to determine whether radiological findings of hemophilic joint disease correlate with serological angiogenic markers. This may enable the development of biomarkers for hemophilic joint disease.

Findings from this study will enable the development of ultrasound as a user friendly tool in the hemophilia clinic in order to understand whether every pain and swelling in a joint is actually a joint bleed or soft tissue bleed and to monitor for joint changes to institute or augment scheduled factor infusions ( prophylaxis). This will also result in significant improvement in quality of life with tailored prophylaxis .

DETAILED DESCRIPTION:
Background: Hemophilic joint disease secondary to recurrent hemarthroses is one of the most disabling and costly complications of hemophilia. Prior to widespread use of prophylactic factor concentrates, children in the United States with severe hemophilia A and B (X-linked recessive disorders with <1% factor VIII/IX (FVIII/FIX) activity) experienced an average of 30-35 hemarthroses per year reported for FVIII deficiency (3,4 ). Clinical and sub clinical hemarthroses during childhood results in synovitis (hypertrophied synovium characterized by villous formation, markedly increased vascularity and chronic inflammatory cells (5) eventually leading to pannus formation and destructive arthritis (6, 7). At this time, synovial bleeding may be related not only to clotting factor deficiency but also to pre-existing vascular damage and inflammation, which is difficult to control clinically. Use of factor concentrate prophylaxis results in hemophilia patients experiencing fewer joint bleeds, less rapid deterioration of joint function and fewer days lost from school or work. However, it may be complicated by the unpredictable development of an inhibitor (a high-affinity, polyclonal, function-neutralizing antibody directed against FVIII/FIX), with an incidence of about 25% and 6% respectively (8) . These individuals have limited treatment options or are treated with products that are less efficacious in treating the joint bleed along with potential deleterious side effects such as thrombogenecity( 9) thus favoring joint disease development.

Primary prophylaxis (infusion of FVIII concentrates (25 - 40 u/kg thrice weekly or FIX concentrates - 80-100u/kg twice a week starting at age 1-2 yrs) before the onset of joint bleeds is used in Sweden since the 1960s to keep the trough level of factor VIII/FIX > 1%, converting a severe hemophilia patient (FVIII/FIX activity <1%) into a milder form (FVIII/FIX >5%) (10 ) . This strategy is expensive (~ $77,760/year for a 20 kg child based on the use of 3000 to 6,000 u/kg/yr with recombinant factor VIII), and may require the use of venous access devices in young children, which is complicated by severe infections, bleeding and thrombosis (11) . Secondary prophylaxis on the other hand, which involves the use of FVIII/FIX concentrates after "target joints" (at least four bleeds occurring into a single joint in the previous six months) have been identified may limit bleeding and subsequent joint damage. However, progression of existing joint disease continues and it is unclear whether secondary prophylaxis can actually prevent joint deterioration (12) . Furthermore, studies comparing primary and secondary prophylaxis in relation to cost-effectiveness and long-term joint morbidity suggest that primary prophylaxis improved long-term joint outcome but was twice as expensive (13 ) . For these reasons, the optimum age, subject population, and timing of prophylaxis is highly debated. Finally, therapeutic options for individuals who fail or cannot use prophylaxis (inhibitor patients) or refuse prophylaxis include isotopic (IS) and surgical synovectomy. Isotopic synovectomy involves intraarticular injection of 32P- colloid with the intent of scarring off the synovium leading to a subsequent reduction in hemarthroses (14) , both procedures being recommended for patients with chronic synovitis and ongoing hemarthroses. Again, the timing of these strategies in relation to the onset of synovitis remain unclear. Hence, if prophylaxis is not started early (before the occurrence of joint bleeds) and subject population is not optimized, a strategy to detect and monitor synovitis and joint arthropathy is urgently needed so that prophylaxis and synovectomy can be timed based on evidence to reap optimum benefits. Furthermore, in hemophilic children who complain of joint pains, clinical examination sometimes, may not clearly define whether the symptoms are related to a joint bleed, synovitis or surrounding soft tissue bleeds. Studies in animals suggest that cartilage damage can occur concurrently with synovial damage (15) contributing to joint arthropathy. Therefore, it seems that determination of both synovial and cartilage changes would be imperative and may help to guide prophylaxis.

Traditionally, hemophilic arthropathy has been diagnosed by clinical examination and plain radiographs of joints, which together tend to underestimate the extent of joint destruction (16) . Magnetic Resonance Imaging (MRI) can estimate the degree of bony damage associated with hemophilic joint disease (14 , 17 -19). The investigators have previously shown the utility of ultrasound-power Doppler sonography( USG-PDS) in detecting synovitis associated with hemophilic joint disease when compared to MRI ( 1) . The need for sedation in children and high costs ($ 2500 for MRI with sedation versus $ 600 for USG- PDS - no sedation at this institution) override the utility of this tool when repeated studies may be required for closer surveillance of joint disease progression. Visualization of cartilage is clinically relevant because benefits of both prophylaxis and synovectomy are realized only if there is minimal damage to cartilage. Furthermore, there is scattered evidence to suggest that isotopic synovectomy in a joint affected by bony arthropathy can lead to progression of the arthropathy leading to crippling arthritis.

The pathogenesis of HJD is not well defined. Neoangiogenesis is a critical factor in processes, such as tumor growth and inflammatory arthritis (20). Increased vascularity and neoangiogenesis have been implicated in the progression of musculoskeletal disorders and tumor growth. Vascular endothelial growth factor (VEGF), the principal signaling molecule in angiogenesis, can be induced by hypoxia and certain cytokines through interaction with its receptors, VEGFR1 and VEGFR2 (21 -23). The synovitic pannus in other joint diseases that share histologic similarities with hemophilic joint disease (HJD) have enhanced oxygen demand and show evidence of de novo blood vessel formation, including endothelialization of the synovium( 24) . Further, VEGF expression in the serum has been correlated with disease activity in rheumatoid arthritis ( 25) . Endothelialization may occur as a result of mature endothelial cell migration or through the recruitment of bone marrow (BM)-derived endothelial progenitor cells (EPCs) and hematopoietic progenitor cells (HPCs) from the peripheral circulation (26) . Importantly, proliferating synovium can secrete chemocytokines, such as VEGF, that might promote recruitment of endothelial cells (ECs) to sites of active angiogenesis ( 25) . Co-localization of hypoxia-inducible factor- 1 (HIF-1 α) which is a transcription factor involved in the induction of VEGF and produced in response to hypoxia within the joint and VEGF emphasizes the role of hypoxia in the up-regulation of angiogenesis in rheumatoid joint diseases ( 27).

The investigators have previously observed a 4-fold elevation in proangiogenic factors (vascular endothelial growth factor-A [VEGF-A], stromal cell-derived factor-1, and matrix metalloprotease-9) and proangiogenic macrophage/monocyte cells (VEGF+/CD68+ and VEGFR1+/CD11b +) in the synovium and peripheral blood of hemophilic joint disease (HJD) subjects along with significantly increased numbers of VEGFR2+/AC133 + endothelial progenitor cells and CD34+/ VEGFR1+ hematopoietic progenitor cells. Sera from HJD subjects induced an angiogenic response in endothelial cells that was abrogated by blocking VEGF, whereas peripheral blood mononuclear cells from HJD subjects stimulated synovial cell proliferation, which was blocked by a humanized anti-VEGF antibody (bevacizumab). Human synovial cells, when incubated with HJD sera, could elicit up-regulation of HIF-1α mRNA with HIF-1α expression in the synovium of HJD subjects, implicating hypoxia in the neoangiogenesis process. The investigators results provided evidence of local and systemic angiogenic response in hemophilic subjects with recurrent hemarthroses suggesting a potential to develop surrogate biologic markers to identify the onset and progression of hemophilic synovitis( 2). Therefore, evidence of increased synovial vascularity on USG-PDS and elevated angiogenic markers suggestive of increased vascularity in hemophilic joint disease subjects provides a compelling opportunity to develop surrogate biological markers for hemophilic joint disease. This would also further aid in tailoring strategies such as prophylaxis and synovectomy in an individual patient.

ELIGIBILITY:
Inclusion Criteria:

1. All children ages 6 months - 18 years with hemophilia A or B
2. Hemophilia subjects with and without a history of hemarthroses including target joints ( joint of interest) and joints without documented bleeds( control joints)
3. Hemophilia subjects with a history of inhibitor to FVIII or FIX and documented hemarthroses
4. History of hemarthroses more than 4 weeks prior to study enrolment to allow for resolution of hemarthroses which could affect detection of synovial and cartilage changes

Exclusion Criteria:

1. Bleeding disorder subjects without a diagnosis of hemophilia
2. Hemophilia subjects with any underlying illness such as liver or renal disease or any systemic illness such as diabetes or any other chronic illness apart from the hemophilia
3. Hemophilia subjects on medications which could increase bleeding risk such as non steroidal anti inflammatory agents, anti seizure medications apart from factor concentrates
4. History of hemarthroses within the 4 weeks prior to study enrolment

Ages: 6 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys with hemophilia and inherited bleeding disorders with and without a history of hemarthroses
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence rates of synovial and cartilage changes using USG-PDS: | 12 months
  Synovial changes on USG- PDS:
  Scoring system for synovitis which has 2 components - joint effusion and synovial thickening: Joint effusion will be defined as a compressible anechoic intracapsular area and the amount of fluid will be semiquantitatively scored usinga previosuly described scoring system by Martinoli et al. Quantitative assessment of the power Doppler signal: Power Doppler signal will be assessed subjectively for degree of vascularity -Table 2, Table 2
  Degree of Vascularity PDS Signal Score Normal or minimal No signal or local dark red 1 Mild hyperemia Dark red to red 2 Moderate hyperemia Red to orange 3 Marked hyperemia Orange to yellow 4

SECONDARY OUTCOMES:
To determine whether the presence/absence of synovial and cartilage changes measured using USG-PDS are associated with any changes in biological surrogate marker levels. | 15 months
  Blood will be collected on the smae day of the study to measure synovial angiogenesis markers- VEGF, MMP-9, SDF-1, HIF-1 , endothelial progenitor cells and hematopoietic progenitor cells

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute of Medical Research Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Acharya SS, Schloss R, Dyke JP, Mintz DN, Christos P, DiMichele DM, Adler RS. Power Doppler sonography in the diagnosis of hemophilic synovitis--a promising tool. J Thromb Haemost. 2008 Dec;6(12):2055-61. doi: 10.1111/j.1538-7836.2008.03160.x. Epub 2008 Sep 23. PMID 18823337
- [Result] Acharya SS, Kaplan RN, Macdonald D, Fabiyi OT, DiMichele D, Lyden D. Neoangiogenesis contributes to the development of hemophilic synovitis. Blood. 2011 Feb 24;117(8):2484-93. doi: 10.1182/blood-2010-05-284653. Epub 2010 Dec 16. PMID 21163925
- [Result] Jansen NW, Roosendaal G, Lundin B, Heijnen L, Mauser-Bunschoten E, Bijlsma JW, Theobald M, Lafeber FP. The combination of the biomarkers urinary C-terminal telopeptide of type II collagen, serum cartilage oligomeric matrix protein, and serum chondroitin sulfate 846 reflects cartilage damage in hemophilic arthropathy. Arthritis Rheum. 2009 Jan;60(1):290-8. doi: 10.1002/art.24184. PMID 19116938
- [Result] Manco-Johnson MJ, Riske B, Kasper CK. Advances in care of children with hemophilia. Semin Thromb Hemost. 2003 Dec;29(6):585-94. doi: 10.1055/s-2004-815626. PMID 14719175
- [Result] Aledort LM, Haschmeyer RH, Pettersson H. A longitudinal study of orthopaedic outcomes for severe factor-VIII-deficient haemophiliacs. The Orthopaedic Outcome Study Group. J Intern Med. 1994 Oct;236(4):391-9. doi: 10.1111/j.1365-2796.1994.tb00815.x. PMID 7931042
- [Result] Madhok R, Bennett D, Sturrock RD, Forbes CD. Mechanisms of joint damage in an experimental model of hemophilic arthritis. Arthritis Rheum. 1988 Sep;31(9):1148-55. doi: 10.1002/art.1780310910. PMID 3048275
- [Result] Ehrenforth S, Kreuz W, Scharrer I, Linde R, Funk M, Gungor T, Krackhardt B, Kornhuber B. Incidence of development of factor VIII and factor IX inhibitors in haemophiliacs. Lancet. 1992 Mar 7;339(8793):594-8. doi: 10.1016/0140-6736(92)90874-3. PMID 1347102
- [Result] Wight J, Paisley S. The epidemiology of inhibitors in haemophilia A: a systematic review. Haemophilia. 2003 Jul;9(4):418-35. doi: 10.1046/j.1365-2516.2003.00780.x. PMID 12828678
- [Result] Lusher JM. Thrombogenicity associated with factor IX complex concentrates. Semin Hematol. 1991 Jul;28(3 Suppl 6):3-5. No abstract available. PMID 1780767
- [Result] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129
- [Result] Blanchette VS, Al-Musa A, Stain AM, Ingram J, Fille RM. Central venous access devices in children with hemophilia: an update. Blood Coagul Fibrinolysis. 1997 Aug;8 Suppl 1:S11-4. PMID 9351530
- [Result] Manco-Johnson MJ, Nuss R, Geraghty S, Funk S, Kilcoyne R. Results of secondary prophylaxis in children with severe hemophilia. Am J Hematol. 1994 Oct;47(2):113-7. doi: 10.1002/ajh.2830470209. PMID 8092125
- [Result] Valentino LA, Hakobyan N, Enockson C, Simpson ML, Kakodkar NC, Cong L, Song X. Exploring the biological basis of haemophilic joint disease: experimental studies. Haemophilia. 2012 May;18(3):310-8. doi: 10.1111/j.1365-2516.2011.02669.x. Epub 2011 Nov 2. PMID 22044636
- [Result] Nuss R, Kilcoyne RF, Geraghty S, Shroyer AL, Rosky JW, Mawhinney S, Wiedel J, Manco-Johnson M. MRI findings in haemophilic joints treated with radiosynoviorthesis with development of an MRI scale of joint damage. Haemophilia. 2000 May;6(3):162-9. doi: 10.1046/j.1365-2516.2000.00383.x. PMID 10792474
- [Result] Lundin B, Manco-Johnson ML, Ignas DM, Moineddin R, Blanchette VS, Dunn AL, Gibikote SV, Keshava SN, Ljung R, Manco-Johnson MJ, Miller SF, Rivard GE, Doria AS; International Prophylaxis Study Group. An MRI scale for assessment of haemophilic arthropathy from the International Prophylaxis Study Group. Haemophilia. 2012 Nov;18(6):962-70. doi: 10.1111/j.1365-2516.2012.02883.x. Epub 2012 Jul 5. PMID 22765835
- [Result] Joseph-Silverstein J, Rifkin DB. Endothelial cell growth factors and the vessel wall. Semin Thromb Hemost. 1987 Oct;13(4):504-13. doi: 10.1055/s-2007-1003526. PMID 3321439
- [Result] Ortega N, Jonca F, Vincent S, Favard C, Ruchoux MM, Plouet J. Systemic activation of the vascular endothelial growth factor receptor KDR/flk-1 selectively triggers endothelial cells with an angiogenic phenotype. Am J Pathol. 1997 Nov;151(5):1215-24. PMID 9358746
- [Result] Maeno N, Takei S, Imanaka H, Takasaki I, Kitajima I, Maruyama I, Matsuo K, Miyata K. Increased circulating vascular endothelial growth factor is correlated with disease activity in polyarticular juvenile rheumatoid arthritis. J Rheumatol. 1999 Oct;26(10):2244-8. PMID 10529148